CLINICAL TRIAL: NCT01288365
Title: Impact of Exercise Training on Functional Capacity in Heart Failure Patients With Preserved Ejection Fraction.
Brief Title: The Impact of Exercise Training on Functional Capacity in Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Clalit Health Services (Other); Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MeirMc K015/2011
Record Dates: First submitted 2011-01-26; First posted 2011-02-02 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: heart failure; preserved ejection fraction
MeSH Terms: conditions — Heart Failure | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise training (Experimental): Protocol of 3 month exercise training program.
  Interventions: Behavioral: Exercise training
- Control (No Intervention): Control group

INTERVENTIONS:
Behavioral: Exercise training — Exercise training program for 3 months (two times a week).
  Arms: Exercise training

SUMMARY:
The purpose of this study is to determine whether exercise training will improve functional capacity in patients with heart failure and preserved ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Clinical heart failure
* Preserved ejection fraction (>50%)
* Stable clinically
* New York Heart Association Class II-III

Exclusion Criteria:

* Unable to exercise
* Other debilitating or unstable disease limiting length of life
* Implanted pacemaker

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of peak oxygen uptake on graded exercise. | After 3 month exercise training
  Changes in physical fitness after 3 month exercise training. This will be measured by a cardiopulmonary exercise test with recording of maximal oxygen uptake during incremental exercise.

SECONDARY OUTCOMES:
Change from baseline of six minute walk | After 3 month exercise training
  Change in the distance covered during a 6 minute walk after 3 month exercise training.
Change from baseline of NYHA class | After 3 month exercise training
  Change in subjective assessment of function capacity based on the New York Heart Association Class classification after 3 month exercise training.

CONTACTS AND LOCATIONS:
Overall Officials: Israel Gotsman, MD, Principal Investigator — Hadassah University Hospital
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel